CLINICAL TRIAL: NCT06605248
Title: NOTUS Feasibility Trial: Enhancing Chronic Back Pain Management With Mobile App-based Pain Education and Clinical Hypnosis in Primary Care
Brief Title: NOTUS Feasibility Study: Reducing Chronic Low Back Pain With Mobile App Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuroscience Research Australia (Other)
Responsible Party: Principal Investigator, James McAuley, Principal Investigator, Neuroscience Research Australia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: X23-0202 & 2023/ETH00540
Record Dates: First submitted 2024-09-10; First posted 2024-09-20 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- App-based self-management tool plus usual care (Experimental): App-based self-management tool consisting of pain education and clinical hypnosis delivered after usual care.
  Interventions: Behavioral: App-based self-management tool plus usual care
- Patient information digital fact-sheet plus usual care (Experimental): The intervention consists of a fact-sheet delivered after usual care.
  Interventions: Behavioral: Patient information digital fact-sheet plus usual care

INTERVENTIONS:
Behavioral: App-based self-management tool plus usual care — The app-based self-management tool will be delivered after patients receive usual care from their general practitioners. The 8-week mobile app intervention will involve daily sessions on pain education and clinical hypnosis for back pain management (5 minutes, 15 minutes of listening to hypnotherapy audio and engaging in physical/social activities for 5 minutes.
  Arms: App-based self-management tool plus usual care
Behavioral: Patient information digital fact-sheet plus usual care — The face-sheet will be delivered after patients receive usual care from their general practitioners.This digital intervention will contain educational material for chronic back pain that includes details about diagnosis, prognosis and treatment options.
  Arms: Patient information digital fact-sheet plus usual care

SUMMARY:
This feasibility study will investigate the feasibility of screening, recruiting, and delivering a mobile app intervention that involves pain education and clinical hypnosis to people seeking treatments for chronic low back pain (chronic LBP) in general practices in Australia.

This study aims to assess the recruitment strategy, the willingness of participants to be included in the proposed treatments, whether the intervention can be delivered as intended within the health care system and clinical setting, the adherence of participants to the proposed treatment, response rates to questionnaires, loss to the short-term follow-up, and the appropriateness and acceptability of the interventions. This feasibility study will inform possible modifications in the recruitment and treatments for the main clinical trial.

A total of 60 participants will be randomised into two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing chronic LBP, defined as pain in the area between the 12th rib and buttock crease accompanied or not by leg pain for a minimum duration of 12 weeks.
* LBP with or without leg pain (in case of leg pain, LBP is worse than leg pain).
* Currently attending general practice across Australia.
* Mean pain intensity score on the NRS ≥ 3/10 in the past week.
* A score of at least moderate on question 8 of the physical functioning component of the SF36 questionnaire.
* Access to a mobile device with minimal requirements to download the study app (300MB).
* Internet connection to access the mobile app functionalities.
* Able to understand English via reading and audio materials.
* Individuals who reported interest in participating in a clinical trial involving digital interventions after consultation with their general practitioners.
* Individuals whose general practitioners permitted them to receive information about the trial after the general practice consultation.

Exclusion Criteria:

* Known or suspected back-specific (e.g., radiculopathy, fracture) or non-back-specific (e.g., tumour, infection) serious spinal pathology.
* Less than six months post-spinal surgery.
* Scheduled for major surgery during the program or the follow-up period.
* Known or suspected serious psychiatric condition not being treated by a health professional that would impact the adherence to the trial activities.
* Known or suspected sight or hearing problems that would limit access to the intervention components (reading and listening using headphones).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
Individuals meeting the preliminary eligibility criteria | From the recruitment start date until the randomisation of 60 participants or 1 year, whichever came first, assessed every week.
  Proportion of individuals meeting the preliminary eligibility criteria in the pre-consultation tool BetterConsult and who agreed to receive a digital intervention as part of the study, compared to all eligible individuals reporting back pain as the primary health issue in the BetterConsult tool (data from BetterConsult).
General practitioners who agreed to prescribe a digital intervention | From the recruitment start date until the randomisation of 60 participants or 1 year, whichever came first, assessed every week.
  Proportion of general practitioners who agreed to prescribe a digital intervention as part of the study compared to all eligible individuals (data from BetterConsult).
Individuals who recieved participant information form compared to those that met the preliminary eligibility criteria | From the recruitment start date until the randomisation of 60 participants or 1 year, whichever came first, assessed every week.
  Proportion of individuals who received the Participant Information Form and shared their name, phone number, and email to be contacted by the research group (data from the research group) compared to those who met the preliminary eligibility criteria and whose general practitioners agreed to prescribe a digital intervention as part of the trial (data from BetterConsult).
Individuals who completed the full eligibility criteria compared to those who shared their details | From the recruitment start date until the randomisation of 60 participants or 1 year, whichever came first, assessed every week.
  Proportion of individuals who completed the full eligibility criteria for the study compared to those who shared their details after receiving the Participant Consent Form (data from the research group).
Number of individuals who provided consent to participate | From the recruitment start date until the randomisation of 60 participants or 1 year, whichever came first, assessed every week.
  Number of individuals who provided consent to participate in the feasibility study (collected by the research group via REDCap).
Number of individuals who provided consent for the research group to collect MBS and PBS data. | From the recruitment start date until the randomisation of 60 participants or 1 year, whichever came first, assessed every week.
  Number of individuals who provided consent for the research group to collect Medicare Benefits Scheme and Pharmaceutical Benefits Scheme data (collected by the research group via REDCap).
Proportion of individuals who completed the baseline questionnaires | From the recruitment start date until the randomisation of 60 participants or 1 year, whichever came first, assessed every week.
  Proportion of individuals who completed the socio-demographic baseline questions compared to all individuals who consented to participate in the feasibility study (data from the research group).
Recruitment rate per day, week or month. | From the recruitment start date until the randomisation of 60 participants or 1 year, whichever came first, assessed every week.
  Number of individuals randomised in a given day, week or month (collected by the research group via REDCap)
The Acceptability of Intervention Measure | Baseline and 8 week follow-up
  The Acceptability of Intervention Measure (AIM) questionnaire ranges from 1 to 5; completely disagree, disagree, neither agree nor disagree, agree, completely agree. Higher scores indicate greater acceptability.
The Appropriateness of Intervention Measure | Baseline and 8 week follow-up
  The Appropriateness of Intervention Measure (AIM) questionnaire ranges from 1 to 5; completely disagree, disagree, neither agree nor disagree, agree, completely agree. Higher score indicates a higher level of appropriateness.
Completion rate of questionnaires | Baseline and 8 week follow-up
  The completion rate of questionnaires at baseline and the eight-week follow-up include: 0 to 10 numeric rating scale average pain and worst pain intensity, 0 to 24 Ronald Morris Disability Questionnaire and DASS-21 (depression, anxiety and stress sub-scales), higher scores indicate worse outcomes. Acceptability of Intervention Measure and Intervention Appropriateness Measure (1 to 5, higher scores indicate better outcomes)
  The completion rate of questionnaires at the 8-week follow-up include: -5 to 5 Global Perceived Effect Scale, 0 to 1 EuroQol 5 dimensions questionnaire, 0 to 12 Short-Form Pain Self-Efficacy Questionnaire, 0 to 100 Credibility/Expectancy Questionnaire (expectancy sub-scale) and 1 to 5 Mobile App Rating Satisfaction Sub-Scale, higher scores indicate better outcomes. 0 to 28 Short-Form Pain Catastrophising Scale, 9 to 45 Back Beliefs Questionnaire, 11 to 44 Short-Form Tampa Scale for Kinesiophobia, higher scores indicate worse outcomes.
Adherence to the digital intervention | Throughout the intervention to the 8 week follow-up
  The proportion of individuals who adhered to the digital intervention (i.e., the proportion of participants who completed each session (data from Mindset Health).
Mobile App Rating Satisfaction Sub-Scale | 8 week follow-up
  We will assess satisfaction sub-scale using two questions from the Mobile App Rating Scale. Each item ranges from 1 to 5 (higher score indicates a greater level of satisfaction).
Participants experience through semi-structured interview | 8 week follow-up
  Qualitative study on participants experience in the feasibility study (with at least 6 participants).
Adverse events | 8 week follow-up
  Assessed by self-reported information
Participants experience with the intervention | 8-week follow-up
  This study will qualitatively investigate the participants experience with three open-ended questions. These questions include: 1. What have you learned or experienced that has been the most helpful to you? 2. How do you see yourself applying the intervention to your daily life in the long term? 3. What else could we do to help you incorporate the intervention into your daily life?

CONTACTS AND LOCATIONS:
Overall Officials: James H McAuley, PhD, Principal Investigator — Neuroscience Research Australia
Locations (1):
- Neuroscience Research Australia, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made to interested researchers only upon reasonable request and once the proposed research project has received separate ethics approval from a Human Research Ethics Committee.
  Request to the data custodian, the Principal Investigator (j.mcauley@neura.edu.au).
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available after the publication of study reports. There is no end date for the availability of study data.
Access Criteria: Protocol and ethics must be provided.